CLINICAL TRIAL: NCT00915902
Title: Fish Oil Treatment for Dyslipidemia Associated With Children and Adolescents
Brief Title: Fish Oil Study for High Triglyceride Levels in Children
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Babu Balagopal (Other)
Collaborators: GlaxoSmithKline (Industry); Johns Hopkins University (Other); Thomas Jefferson University (Other)
Responsible Party: Sponsor-Investigator, Babu Balagopal, Principal Research Scientist, Nemours Children's Clinic
Organization: Nemours Children's Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: GIDDING
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Omacor; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3-acid ethyl esters (Lovaza) (Experimental): This randomized, double-blind, placebo, crossover trial consisted of two 8-week treatment periods, separated by a 4-week washout. Eligible patients were randomized to receive either fish oil 4 g daily or corn oil placebo during the first 8-week treatment period; patients received the alternate treatment during the next treatment period. GlaxoSmithKline supplied the study drug and the placebo. The study drug, Omega-3-acid ethyl esters (Lovaza) was given to patients PO daily as two, 1 g capsules taken twice daily during the duration of their 8-week treatment period. The study drug contained minimally 1.5 g DHA (docosahexaenoic acid) and 1.86 g EPA (eicosapentaenoic acid).
  Interventions: Drug: Omega-3-acid ethyl esters
- Placebo (Placebo Comparator): This randomized, double-blind, placebo, crossover trial consisted of two 8-week treatment periods, separated by a 4-week washout. Eligible patients were randomized to receive either fish oil 4 g daily or corn oil placebo during the first 8-week treatment period; patients received the alternate treatment during the next treatment period. The corn oil placebo was given to patients PO daily as two, 1 g capsules taken twice daily during the duration of their 8-week non-treatment (placebo) period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega-3-acid ethyl esters — Omega-3-acid ethyl esters (Lovaza), two 1-gram capsules taken twice daily for 8 weeks
  Other Names: Lovaza
  Arms: Omega-3-acid ethyl esters (Lovaza)
Drug: Placebo — Placebo (corn oil), two 1-gram capsules taken twice daily for 8 weeks
  Other Names: Corn Oil
  Arms: Placebo

SUMMARY:
High triglyceride levels are increasingly recognized in children, particularly those who are overweight. There are no studies of treatment of high triglycerides in children and adolescents. Fish oil is attractive because it is considered safe and effective for treating high triglycerides in adults and has been used safely for other purposes in children. The investigators will conduct a randomized study of Lovaza (the only prescription omega-3 fish oil medication) in 44 children and adolescents to study efficacy in lowering triglycerides, safety, and possible mechanisms of beneficial effects.

DETAILED DESCRIPTION:
Participants (n = 42, age 14 + 2 yrs) with hypertriglyceridemia and LDL cholesterol < 160 mg/dl were enrolled in a randomized double blind cross over trial comparing 4 g fish oil daily with placebo. Treatment interval was 8 weeks with a 4 week wash out, between the two treatment intervals. Lipid profile, lipoprotein particle distribution and size, glucose, insulin, high sensitivity C reactive protien (CRP), interleukin-6, fibrinogen, plasminogen activator inhibitor-1 (PAI-1), and thrombin generation were measured.

Patients were evaluated at 6 time points: Visit 1/baseline (week 0), Visit 2/randomization (week 4), Visit 3/after treatment 1 (week 12) , Visit 4/after wash out (week 16), Visit 5/after treatment 2 (week 24) and Visit 6/close out (week 28) . Patients were advised to maintain a stable diet and not alter baseline fish consumption . One participant took an oral contraceptive throughout the trial. Any fish oil supplements were discontinued. Advice on a heart healthy diet was provided. Blood pressure (right arm sitting with appropriate sized cuff, taken 3 times, last measurement used), height, and weight were measured at the beginning of the study, after the first wash out period, and close out. Participant phone contact was made during each treatment arm to assess diet stability. Fasting lipid profile was performed at every visit. Red blood cell fatty acid profile and secondary endpoints were performed at all visits except baseline.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who are 10-17 years of age
* Fasting triglyceride level >150 mg/dl and < 750 mg/dl measured on 2 separate occasions.
* Ability to follow the study procedures and adhere to the diet counseling recommendations
* Written parental permission and assent are obtained prior to any research procedures

Exclusion Criteria:

* Bleeding disorders
* Diabetes mellitus (impaired glucose tolerance is not an exclusion)
* Uncontrolled hypothyroidism
* Liver disease
* Allergy to fish/shellfish
* Patients requiring chronic use of aspirin and non-steroidal anti-inflammatory agents
* Patients requiring lipid lowering agents
* LDL-Cholesterol levels >160 mg/dl
* Current participation in another clinical study or within the previous 30 days
* Alcohol use
* Currently pregnant or planning to become pregnant during the course of this trial (confirmed by pregnancy testing)
* Any significant medical condition which the investigator believes would interfere with the patient's ability to safely participate in this trial

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2009-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Gidding, MD, Principal Investigator — Nemours
Locations (3):
- United States (3):
  - A. I. duPont Hospital for Children, Wilmington, Delaware
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Thomas Jefferon University, Philadelphia, Pennsylvania

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Nemours Alfred I. duPont Hospital for Children, Johns Hopkins University and Thomas Jefferson University. Recruitment took place between July 2009 and December 2011.
Pre-assignment Details: Patients completed a 4 week dietary run-in prior to randomization at visit 2.
Groups:
- Lovaza Then Placebo: Omega-3-acid ethyl esters (Lovaza) two 1-gram capsules taken twice daily for 8 weeks, then 4 week washout, then Placebo for 8 weeks
- Placebo Then Lovaza: Placebo for 8 weeks, then 4 week washout, then Omega-3-acid ethyl esters (Lovaza) two 1-gram capsules taken twice daily for 8 weeks
Period: 1st Treatment Period
Arm/Group | Lovaza Then Placebo | Placebo Then Lovaza
Started | 20 | 22
Completed | 19 | 22
Not Completed | 1 | 0
Period: Washout (4 Weeks)
Arm/Group | Lovaza Then Placebo | Placebo Then Lovaza
Started | 19 | 22
Completed | 19 | 21
Not Completed | 0 | 1
Period: 2nd Treatment Period
Arm/Group | Lovaza Then Placebo | Placebo Then Lovaza
Started | 19 | 21
Completed | 19 | 20
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Lovaza) Followed by Placebo: Omega-3-acid ethyl esters (Lovaza) two 1-gram capsules taken twice daily for 8 weeks followed by placebo for 8 weeks
- Placebo Followed by Treatment (Lovaza): Placebo, two 1-gram capsules (corn oil) taken twice daily for 8 weeks followed by treatment (Lovaza) for 8 weeks
- Total: Total of all reporting groups
Arm/Group | Treatment (Lovaza) Followed by Placebo | Placebo Followed by Treatment (Lovaza) | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (0.4) | 14.2 (0.5) | 14.1 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 8 | 13
  Male | 15 | 14 | 29
Region of Enrollment [Number; unit: participants]
  United States | 20 | 22 | 42
Triglyceride (mg/dL [Mean (Standard Deviation); unit: mg/dL] | 260 (22) | 280 (25) | 270 (24)

OUTCOME MEASURES:

1. Primary Outcome: Change in Triglyceride Level
Time Frame: after 8 week treatment or placebo period
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- Omega-3-acid Ethyl Esters (Lovaza): Omega-3-acid ethyl esters: Omega-3-acid ethyl esters (Lovaza) two 1-gram capsules taken twice daily
- Placebo: Placebo: Placebo, two 1-gram capsules taken twice daily for 8 weeks
Arm/Group | Omega-3-acid Ethyl Esters (Lovaza) | Placebo
Number analyzed (Participants) | 39 | 39
mg/dL | -52 (16) | -16 (15)

ADVERSE EVENTS:
Time Frame: During the 20 week duration of the clinical trial. Specifically, during the first 8 week treatment period, the subsequent 4 week washout period, and the following 8 week treatment period.
Description: Adverse Events were only collected and reported during the clinical trial, not after the conclusion of the trial, or prior to its start.
Groups:
- Treatment (Lovaza) Followed by Placebo, During Treatment: Omega-3-acid ethyl esters (Lovaza) two 1-gram capsules taken twice daily for 8 weeks followed by placebo for 8 weeks. Adverse events during 8 weeks of treatment before placebo.
- Treatment (Lovaza) Followed by Placebo, During Placebo: Omega-3-acid ethyl esters (Lovaza) two 1-gram capsules taken twice daily for 8 weeks followed by placebo for 8 weeks. Adverse events during 8 weeks of placebo, after 8 weeks of treatment and 4 weeks of washout.
- Placebo Followed by Treatment (Lovaza), During Placebo: Placebo, two 1-gram capsules (corn oil) taken twice daily for 8 weeks followed by 4 week washout then treatment (Lovaza) for 8 weeks. Adverse events during 8 week placebo, after 8 weeks of treatment with Lovaza and a 4 week washout.
- Placebo Followed by Treatment (Lovaza), During Treatment: Placebo, two 1-gram capsules (corn oil) taken twice daily for 8 weeks followed by 4 week washout then treatment (Lovaza) for 8 weeks. Adverse events during 8 week Treatment with Lovaza that followed 8 weeks of placebo and a 4 week washout.
Arm/Group | Treatment (Lovaza) Followed by Placebo, During Treatment | Treatment (Lovaza) Followed by Placebo, During Placebo | Placebo Followed by Treatment (Lovaza), During Placebo | Placebo Followed by Treatment (Lovaza), During Treatment
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/22 | 1/22
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/22 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Lovaza) Followed by Placebo, During Treatment (N=20) | Treatment (Lovaza) Followed by Placebo, During Placebo (N=20) | Placebo Followed by Treatment (Lovaza), During Placebo (N=22) | Placebo Followed by Treatment (Lovaza), During Treatment (N=22)
depression, worsening (Psychiatric disorders) | 0 | 0 | 0 | 1 — hospital stay for depression, worsening. not related to study.

LIMITATIONS AND CAVEATS:
Intrinsic variability of triglycerides is large and may have confounded analyses; 4-week washout between treatment periods may have been too short; a reduction of triglycerides in the corn oil placebo group may have compromised the results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No